CLINICAL TRIAL: NCT05758168
Title: Aesthetic Outcome of Tie-over Bolster Application in Surgical Wounds: a Randomized Evaluator-blinded Split-wound Comparative Effectiveness Trial.
Brief Title: Aesthetic Outcome of Tie-over Bolster Application in Surgical Wounds
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Other
Other Study IDs: 1977459
Record Dates: First submitted 2023-02-24; First posted 2023-03-07 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Scarring
Keywords: Tie-over Bolster
MeSH Terms: conditions — Cicatrix

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Two blinded observers will record their scores independently using the POSAS instrument.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Layered Closure (No Intervention): A cutaneous layer of sutures will be placed on one side of wound, as is standard of care.
- Layered Closure with Tie-Over Bolster Dressing (Experimental): The other side of wound will have a cutaneous layer of sutures with the addition of a bolster dressing.
  Interventions: Procedure: Addition of Tie-Over Bolster Dressing

INTERVENTIONS:
Procedure: Addition of Tie-Over Bolster Dressing — Bolster will be sutured into place using peripheral non-absorbable anchoring sutures.
  Arms: Layered Closure with Tie-Over Bolster Dressing

SUMMARY:
When patients have surgery on the head and face, stitches are the standard way to close the wound. Wounds always result in a scar, but doctors are always looking for ways to reduce scarring. Several studies have been done to test ways to close wounds that reduce scarring. One idea is to reduce the tension around the cut. One way to reduce tension is to stitch a small piece of a special gauze over the top of the regular stitches. This procedure is called a "tie-over bolster dressing." As the name implies, this extra dressing "bolsters" the wound closure so that the skin on each side of the cut stays in place.

The bolster dressing procedure has been used in the past in special cases, such as when skin grafts are necessary. The bolster dressing helps the skin graft heal by making sure the graft stays exactly in place. Keeping the wound stable with a bolster dressing also reduces bleeding under the wound. For non-grafted wounds, the bolster dressing procedure has not normally been used, and has not been well-studied. In this study the whole wound will be stitched normally and then the bolster dressing will be applied over half of the wound. This will allow us to see if the side with the bolster dressing heals with less scarring.

DETAILED DESCRIPTION:
Following cutaneous surgical procedures, scar formation is inevitable. Reducing the degree of scar formation and achieving the best aesthetic outcome remains prominent within the dermatological literature. Recent research has highlighted the impact of mechanical forces and tension on scar formation, demonstrating that reducing the mechanical stress within the wound environment results in better aesthetic outcome (1,2). Tension-shielding devices have shown promise in scar reduction in both humans and porcine models (2). More recently, two clinical trials have shown that the use of an "embrace" device, a silicone-based dressing designed to minimize wound tension, effectively improves the aesthetic outcome following scar revision surgery (3,4). In addition, application of negative pressure via vacuum sealing drainage (VSD), commonly called a "wound-vac", has been consistently shown to accelerate wound healing (5). However, using these methods can be challenging, particularly due to cost, practicability, and patient compliance.

An alternative method for reducing mechanical stressors along scars has long been used within dermatologic surgery, namely the application of a bolster dressing.

For decades, tie-over bolster dressings have been employed following cutaneous procedures repaired with skin grafting. Typically, these bolsters are composed of Xeroform gauze (bismuth tribromophenate petrolatum-impregnated gauze) which are sutured on top of the graft. These have been shown to stabilize the graft, immobilize the wound bed, and reduce hematoma formation by delivering persistent downward pressure (6,7).

To our knowledge, the impact of scar cosmesis and rate of post-operative complications following the administration of tie-over bolster dressing over primary linear repair of surgical wounds have not been studied. This study seeks to determine the effectiveness of a tie-over bolster dressing in reducing tension to improve scar cosmesis by using individuals as their own controls in a split-scar model.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Able to give informed consent themselves
* Patient scheduled for cutaneous surgical procedure on the head or neck with predicted primary closure
* Willing to return for follow-up visit

Exclusion Criteria:

* Incarceration
* Under 18 years of age
* Pregnant women
* Unable to understand written and oral English Wounds with predicted closure length less than 3cm

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-10-10 (Actual); Primary Completion 2026-02-25 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Observer Scar Assessment as measured by Patient Observer Scar Assessment Score (POSAS) | 3 months
  The primary endpoint will be the score of two blinded reviewers independently using the POSAS assessment. The observer scale of the POSAS consists of six items (vascularity, pigmentation, thickness, relief, pliability, and surface area). All items are scored on a scale ranging from 1 ("like normal skin") to 10 ("worst scar imaginable"). The sum of the six items results in a total score of the POSAS observer scale. Furthermore, an overall opinion is scored on a scale ranging from 1 to 10. All parameters should preferably be compared to normal skin on a comparable anatomic location.

SECONDARY OUTCOMES:
Patient Scar Assessment as measured by Patient Observer Scar Assessment Score (POSAS) | 3 months
  This is the patient portion of the POSAS assessment, which will be independently recorded. The patient scale of the POSAS consists of six items (pain, itch, thickness, color, stiffness, and irregularity). All items are scored on a scale ranging from 1 ("as normal skin") to 10 ("yes, very different"). The sum of the six items results in a total score of the POSAS patient scale. Furthermore, an overall opinion is scored on a scale ranging from 1 to 10.
Width of Scar as measured using Trace-to-Tape Method | 3 months
  The trace-to-tape method is an objective measure for linear postoperative scars. The mean scar width will be determined using the trace-to-tape method. The surface area of the scar will be collected by tracing the scar with a water-based gel pen. While still wet, the gel residue will be lifted from the skin with clear packing tape and transferred on a sheet of paper.
Complications or Adverse Events from Treatment | 3 months
  For example, if one half of the scar has more associated erythema, as measured using the Trace-to-Tape method, then it will be recorded. Other complications from the treatment will also be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Eisen, MD, Principal Investigator — University of California, Davis - Dermatology
Locations (1):
- University of California, Davis - Dermatology Department, Sacramento, California, United States

REFERENCES:
- [Background] Gurtner GC, Dauskardt RH, Wong VW, Bhatt KA, Wu K, Vial IN, Padois K, Korman JM, Longaker MT. Improving cutaneous scar formation by controlling the mechanical environment: large animal and phase I studies. Ann Surg. 2011 Aug;254(2):217-25. doi: 10.1097/SLA.0b013e318220b159. PMID 21606834
- [Background] Barnes LA, Marshall CD, Leavitt T, Hu MS, Moore AL, Gonzalez JG, Longaker MT, Gurtner GC. Mechanical Forces in Cutaneous Wound Healing: Emerging Therapies to Minimize Scar Formation. Adv Wound Care (New Rochelle). 2018 Feb 1;7(2):47-56. doi: 10.1089/wound.2016.0709. PMID 29392093
- [Background] Longaker MT, Rohrich RJ, Greenberg L, Furnas H, Wald R, Bansal V, Seify H, Tran A, Weston J, Korman JM, Chan R, Kaufman D, Dev VR, Mele JA, Januszyk M, Cowley C, McLaughlin P, Beasley B, Gurtner GC. A randomized controlled trial of the embrace advanced scar therapy device to reduce incisional scar formation. Plast Reconstr Surg. 2014 Sep;134(3):536-546. doi: 10.1097/PRS.0000000000000417. PMID 24804638
- [Background] Lim AF, Weintraub J, Kaplan EN, Januszyk M, Cowley C, McLaughlin P, Beasley B, Gurtner GC, Longaker MT. The embrace device significantly decreases scarring following scar revision surgery in a randomized controlled trial. Plast Reconstr Surg. 2014 Feb;133(2):398-405. doi: 10.1097/01.prs.0000436526.64046.d0. PMID 24105084
- [Background] Liu J, Hu F, Tang J, Tang S, Xia K, Wu S, Yin C, Wang S, He Q, Xie H, Zhou J. Homemade-device-induced negative pressure promotes wound healing more efficiently than VSD-induced positive pressure by regulating inflammation, proliferation and remodeling. Int J Mol Med. 2017 Apr;39(4):879-888. doi: 10.3892/ijmm.2017.2919. Epub 2017 Mar 13. PMID 28290607
- [Background] Seymour FK, Giele HP. Tie-overs under pressure. Br J Plast Surg. 2003 Jul;56(5):494-7. doi: 10.1016/s0007-1226(03)00131-0. PMID 12890464
- [Background] Saikaly SK, Saikaly LE, Steadmon MJ. The use of a horizontal mattress suture and notches in 3% bismuth tribromophenate-impregnated petrolatum gauze tie-over bolster dressings to improve surgical outcomes after skin grafts. J Am Acad Dermatol. 2020 Nov;83(5):e335-e336. doi: 10.1016/j.jaad.2019.06.040. Epub 2019 Jun 25. No abstract available. PMID 31251960